CLINICAL TRIAL: NCT05816616
Title: Pilot Study of Hyperpolarized Xenon Functional Lung Imaging in COPD Patients Undergoing Targeted Lung Denervation
Brief Title: Hyperpolarized Xenon Functional Lung Imaging in COPD Patients Undergoing Targeted Lung Denervation
Status: Withdrawn | Type: Observational
Why Stopped: Did not received funding and it was not started.
Sponsor: Xemed LLC (Industry)
Collaborators: Temple University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 851758
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-01

CONDITIONS: COPD
Keywords: hyperpolarized xenon-129 MRI; COPD; Targeted Lung Denervation (TLD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD-TLD patients: COPD patients to be treated with Targeted Lung Denervation and enrolled in Airflow-3 clinical trial at Temple University Hospital, and which are also willing to participate in hyperpolarized xenon imaging of their lungs prior and poste TLD treatment.
  Interventions: Diagnostic Test: Functional imaging of the lungs using MagniXene (hyperpolarized xenon-129) MRI

INTERVENTIONS:
Diagnostic Test: Functional imaging of the lungs using MagniXene (hyperpolarized xenon-129) MRI — Patients for this observational study will be selected on a voluntarily basis from the ongoing Airflow-3 interventional clinical trial at Temple University Hospital. For this observational sub-study, patients will have their lung function measured using hyperpolarized xenon-129 MRI prior to TLD treatment, and 90 days post-treatment for a better understanding of treatment effects. This sub-study does not influence in any way the patient treatment or the outcomes for the main Airflow-3 TLD clinical trial.

SUMMARY:
Targeted Lung Denervation (TLD) Therapy is intended to improve airway smooth muscle relaxation from the site of treatment all the way to the lung periphery, which may be beneficial in the treatment of patients with COPD. To better understand the physiological effects of this therapy, the investigators intend to conduct a functional magnetic resonance imaging study of the lung with HP 129Xe study in COPD patients undergoing this procedure. HP 129Xe provides valuable regional information about ventilation and gas exchange in both healthy and diseased lung.

DETAILED DESCRIPTION:
This study will be assessing the treatment response using HP 129Xe MRI for patients undergoing Target Lung Denervation (TLD) in COPD patients. Subjects eligible to participate in this study are those who agree and have already consented to participate in the AIRFLOW-3 clinical trial for TLD treatment at Temple University Hospital. The intent of this study is to image lung function using HP 129Xe MRI in ten TLD subjects before and approximately three months post TLD procedure as an observational sub-study. Subjects willing to participate in this sub-study will have to consent to this study and plan for two MRI imaging sessions: one prior TLD and a follow-up at approximately three months post TLD procedure.

As part of this companion protocol at Penn, the aim is to image each subject twice, using a total of 2.5L of HP 129Xe gas administered over approximately 50 breaths during each visit. Using the dynamic image set acquired, the investigators will characterize each imaging voxel (approximately 4mm x 4mm x 4mm) in terms of its tidal volume (in mm3), functional residual capacity (in mm3), fractional ventilation (efficiency of gas exchange via ventilation, unit less), and what is defined as "arrival time", which can be also shown as 'tidal volume hysteresis', and corresponds to the area enclosed when the local tidal volume is plotted against the inhaled gas volume. The latter parameter is zero in a region that inflates and deflates perfectly in sync with the inhaled gas volume but grows in magnitude when the two are out of sync: e.g., in cases obstructed ventilation or air trapping. The subject will be coached to maintain a reasonably steady breathing cadence of 10-15 breaths per minute, depending on their size and natural breathing rate, but will be otherwise unconstrained with respect to breath timing and volume. Each imaging session will take approximately 30 minutes, including positioning in the MRI and inhalation of a small HP 129Xe dose for scanner calibration. The proposed dynamic HP 129Xe MRI technique allows for the quantification of fractional ventilation (FV), tidal volume (TV), functional residual capacity (FRC), arrival time (τ), apparent diffusion coefficient (ADC), and dissolved phase HP 129Xe information. Obtaining all of these parameters in a single scan session reduces the necessary amount of imaging gas while increasing accuracy by correcting artifacts associated with collateral ventilation and the slow filling of parenchyma in diseased lungs. Following the two imaging sessions, data will be analyzed and compared, including comparison with other lung function measuring techniques.

ELIGIBILITY:
Inclusion Criteria:

- Subjects are already consented and enrolled in the AIRFLOW-3 clinical trial at Temple University Hospital and are willing to participate in this sub-study for assessing functional lung changes from prior to post TLD treatment using hyperpolarized xenon-129 MRI.

Exclusion Criteria:

* Patients less than 18 years old;
* Patients known to be pregnant - a positive pregnancy test will be used to respectively exclude pregnant patients;
* Any known contraindication to MRI examination;
* Anyone with an implanted metal device;
* Inability to provide informed consent;
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed participation in the study;
* History of uncompensated organ failure (i.e. organ failure that is not stabilized through medical intervention), which will be assessed by the PI;
* Homelessness or other unstable living situation;
* Active drug or alcohol dependence;
* Claustrophobia;
* Subjects with a BMI>35;
* Subjects with chest size larger than the bore of MRI machine from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the pool of patients with severe COPD enrolled in Targeted Lung Denervation therapy AIFLOW-3 clinical trial ongoing at Temple University Hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in regional lung ventilation from pre-TLD baseline to three months post-TLD. | 3-month
  Fractional ventilation (FV) is defined as the ratio of inspired gas to residual gas volume and it will be measured using dynamic HP 129Xe MRI performed over approximately 50 breaths during normal respiratory cycle in which small amounts of xenon will be precisely administered. FV provides a quantitative and non-dimensional map of inhaled gas within the lungs and it is the most widely accepted quanititative measure of regional lung ventilation. The pre and post measurements will be entered into a general linear model to search for differences.